CLINICAL TRIAL: NCT05790031
Title: Development of Intelligent Nighttime Brace With Smart Padding to Treat of Adolescent Idiopathic Scoliosis
Brief Title: Trials of Intelligent Nighttime Brace With Smart Padding to Treat of Adolescent Idiopathic Scoliosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Joanne Yip, Professor, The Hong Kong Polytechnic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITS/007/22
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Scoliosis, Bracing Treatment
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intelligent Nighttime Brace (Experimental): The design of intelligent nighttime brace will incorporate different mechanism, such as a) compression and pulling forces through a customisable rigid brace, b) lumbar flexion by using a supporting air-belt, c) three-point pressure system is used to exert corrective forces by the intelligent paddings in the transverse direction, d) adjust the pressure of the brace padding through a pressure monitoring system in accordance with the sleeping posture of the users
  Interventions: Device: Intelligent Nighttime Brace

INTERVENTIONS:
Device: Intelligent Nighttime Brace — Participants will be invited to undergo a fitting session of intelligent nighttime brace. After the fitting, participants will join a 6-month wear trial of the intelligent nighttime brace. Participants are required to wear the intelligent nighttime brace for 8 hours a day during sleeping and compliance will be recorded by an intelligent monitoring system. Participants will be invited to undergo assessments before the wear trial, after the trials of 3 months and after the trial of 6 months. The measure outcomes of the assessment include 1)ultrasound scanning image, 2)3D body scanning, 3)garment pressure, 4) questionnaires

SUMMARY:
Adolescent idiopathic scoliosis (AIS) is a three-dimensional spinal deformity usually associated with intervertebral rotation that takes place during adolescence. Generally, bracing treatment is a common option for scoliosis patients. Non-surgical treatment for scoliosis patients is to offer a conservative solution to treat their condition and encourage a higher degree of compliance by avoiding interference with their daily life activities. Therefore, intelligent nighttime braces have been developed to solve this issue, which are intended to be worn for inhibiting the advancement of spinal deformity during sleeping hours. However, its efficacy is still controversial. Intelligent nighttime brace with a specialized design for teenagers with scoliosis is limited and most part of them are lack of mobility and lack of control over corrective forces on particular regions of the vertebra. A scientific approach should be used to design and develop intelligent nighttime brace as a treatment option for adolescents with early scoliosis.

DETAILED DESCRIPTION:
The design of intelligent nighttime brace with smart padding for adolescent idiopathic scoliosis will incorporate different mechanisms, such as

1. compression and pulling forces through a customizable rigid brace
2. lumbar flexion by using a supporting air-belt.
3. three-point pressure system is used to exert corrective forces by the intelligent paddings in the transverse direction
4. adjust the pressure of the brace padding through a pressure monitoring system in accordance with the sleeping posture of the users

ELIGIBILITY:
Inclusion Criteria:

1. between the ages of 10-13,
2. scoliosis with a Cobb angle larger between 10 -25 degrees;
3. No prior treatment
4. Pre-menarche or post- menarche by no more than 1 year
5. Ability to read and understand English or Chinese
6. Physical and mental ability to adhere to intelligent nighttime braces protocol

Exclusion Criteria:

1. History of previous surgical or orthotic treatment for AIS
2. Diagnosis of other musculoskeletal or developmental illness that might be responsible for the spinal curvature
3. Contraindications for pulmonary and/ or exercise tests
4. Psychiatric disorders
5. Recent trauma

Ages: 10 Years to 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Investigate the in-brace Cobb angle | 2 hours and 6 months after wearing the brace
  1. Number of Participants Maintaining Cobb Angle Stability (<5° Increase) After Wearing the Brace for 2 Hours, as Measured by Spine X-ray (AP View).

SECONDARY OUTCOMES:
Contour control | 6 months
  Use a 3D body scanner to measure the contour asymmetry. By using 3D scanning images, the contour asymmetry changes over a six-month period will be assessed.
Force measurements and monitoring | 6 months
  Measure the brace interface pressure by the Novel Pliance-xf-16 analyser. The bio-mechanics of the intelligent nighttime brace are assessed by the changes of the pressure distribution. A real-time intelligent system is use to monitor the pressure distribution.
Health-related quality of life (SRS-22) | 6 months
  Measure the quality of life by validated questionnaire, Euroqol (EQ-5D-5L). The five dimensions of the descriptive system are mobility, self-care, regular activities, pain/comfort, and anxiety/depression. The patients with higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Yip, phd, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, China